CLINICAL TRIAL: NCT03106857
Title: A Proposed Physical Activity and Diet Control to Manage Constipation in Middle Age Obese Women
Brief Title: Effect of Weight Reduction on Constipation
Acronym: constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Associate Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T. REC/012/001535
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Group A (Placebo Comparator): Physical activity, a low caloric diet, and the routine standard care for constipation
  Interventions: Other: Group A
- Group B (No Intervention): No intervention

INTERVENTIONS:
Other: Group A — Group A Physical activity and low caloric diet for
  Arms: Group A

SUMMARY:
In total, 125 women aged between 20 and 40 years were recruited in this study. Participants were considered eligible when they met the inclusion criteria of being diagnosed with functional constipation, as defined by the Rome Foundation. The study was a randomized controlled trial carried out at Cairo University Hospital.Patients whose BMI exceeded 30 kg/m2 were included. In addition, they fulfilled the ROM criteria of constipation.

DETAILED DESCRIPTION:
In total, 125 women aged between 20 and 40 years were recruited in this study. Participants were considered eligible when they met the inclusion criteria of being diagnosed with functional constipation, as defined by the Rome Foundation. The study was a randomized controlled trial carried out at Cairo University Hospital.

Patients whose BMI exceeded 30 kg/m2 were included. In addition, they fulfilled the ROM criteria of constipation, as follows: (1) Suffered from any 2 or more of the following symptoms in the past 12 weeks (not necessarily consecutive), with the onset of symptoms at least 6 months prior to diagnosis: a) straining during at least 25% of defecations, b) lumpy or hard stools in at least 25% of defecations, c) sensation of incomplete evacuation for at least 25% of defecations, d) sensation of anorectal obstruction/blockage for at least 25% of defecations, e) requirement of manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor muscles), and f) fewer than 3 defecations per week; (2) Loose stools rarely occurred without the use of laxatives; (3) Insufficient criteria for irritable bowel syndrome; and (4) Women were sedentary (less than 1 hour/week of physical activity), with no evidence of participation in diet control/weight reduction programs within the last 6 months.

Patients with metabolic, endocrine, and neurologic constipation; current or past smokers; those with any orthopedic limitation; and those with congenital megacolon, pseudo-obstruction, and anorectal disorders were excluded from the study. Patients suffering from constipation due to drugs, disabled patients, and those who had undergone any abdominal surgery during the intervention or those who failed to complete the study protocol were also excluded. All participants provided a written informed consent before enrolling in the study.

Study design and intervention:

Participants were randomly divided into 2 groups. Group A included 62 women who were following a suggested protocol of physical activity and a low caloric diet in addition to the routine standard care for constipation. The low caloric diet allowed 1000-1200 kcal/day, divided as follows: 50%-60% carbohydrates, 20% protein, <30% total fat, and 18 g of fiber /1000 Kcal. The diet plans were revised every 2 weeks and the diet was modified while ensuring that it was within the allowed caloric value, in addition to the routine standard care for constipation. Group B included 63 patients who received only the standard medical care for constipation and a low caloric diet as in Group A. Patients in both groups followed their program for 12 weeks.

Exercise intervention for Group (A) Each woman in Group A participated in the exercise training program for 12 weeks, 3 times per week, with each exercise session lasting for 60 minutes. The participants were instructed not to eat for 3 hours before the exercise session.

The exercise training program was in the form of walking on a treadmill without tightly grasping the rails, because this action seemed to reduce the workload during any stage of the exercise. To overcome this issue, the participants were asked to remove their hands from the rails, close their fists, and place only 1 finger on the rails to maintain balance once they were accustomed to walking on the treadmill.

The exercise session was started by a 10-minute warm-up, which involved walking without any resistance or inclination on the walkway of the treadmill, followed by 40 minutes of walking with 15 degrees of inclination and a speed adjusted to reach 20%-40% of the target heart rate (THR) in the first 6 weeks of the study; the speed was increased to reach 40%-60% THR in the next 6 weeks of the study. The session ended by 10 minutes of recovery period, in which the intensity of the exercise was reduced to the level of the warm-up.

The assessment procedures performed before and after 12 weeks of intervention consisted of the following:

1. The Patient Assessment of Constipation - Symptom (PAC-SYM) is a reliable and valid 16, 17 tool to measure the patient's perspective of constipation symptoms in terms of the frequency and severity. It is a 12-item self-reported measure, which is divided into 3 manifestation subscales (i.e. abdominal, rectal, and stool). Items are scored on a 4-point Likert scale, with a score of 4 demonstrating the worst symptom severity 18, 19.
2. The Patient Assessment of Constipation Quality of Life (PAC-QOL) is a comprehensive measure of the constipation burden on the patient's quality of life (QoL) in terms of functions, activities, and well-being. It is considered a valid and reproducible tool with high internal consistency 20.
3. The Short Form-36 (SF-36) is well validated, reliable, does not require more time or effort to be completed, and has been presented in several international studies 21- 23. It is a 36-item questionnaire that measures the QoL across 8 scales (domains), which are based on both physical and emotional aspects. The 8 domains of SF36 are concerned with the following: physical functioning, role limitations owing to physical health or emotional problems, energy/fatigue, emotional wellbeing, social functioning, pain, and general health. In addition, a single item is included to identify any perceived change in health, making the SF-36 a useful indicator for change in QoL over time and treatment. The scores of the SF-36TM physical component summary and SF-36TM mental component summary are calculated by simply calculating the mean score of all of the physically and emotionally relevant items 23- 25.

Descriptive statistics were calculated as the mean and standard deviation. Inferential statistics evaluated the changes in constipation symptoms, QoL questionnaires, and BMI using unpaired t-test between the 2 groups, while paired t-test was used to measure the changes within a group. Pearson correlation coefficient was used to measure the strength and direction of the relationship between BMI and PAC-SYM scores, and between BMI and QoL. All data were analyzed using SPSS version 18.0 (SPSS, Chicago, IL, USA), with statistical significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients whose BMI exceeded 30 kg/m2 were included.

In addition, they fulfilled the ROM criteria of constipation, as follows:

1. Suffered from any 2 or more of the following symptoms in the past 12 weeks (not necessarily consecutive), with the onset of symptoms at least 6 months prior to diagnosis:

   1. straining during at least 25% of defecations,
   2. lumpy or hard stools in at least 25% of defecations,
   3. sensation of incomplete evacuation for at least 25% of defecations,
   4. sensation of anorectal obstruction/blockage for at least 25% of defecations,
   5. requirement of manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor muscles), and
   6. fewer than 3 defecations per week;
2. Loose stools rarely occurred without the use of laxatives;
3. Insufficient criteria for irritable bowel syndrome; and
4. Women were sedentary (less than 1 hour/week of physical activity), with no evidence of participation in diet control/weight reduction programs within the last 6 months.

Exclusion Criteria:

* Patients with metabolic, endocrine, and neurologic constipation;
* current or past smokers;
* those with any orthopedic limitation; and
* those with congenital megacolon, pseudo-obstruction, and anorectal disorders were excluded from the study.

Patients suffering from constipation due to drugs, disabled patients, and those who had undergone any abdominal surgery during the intervention or those who failed to complete the study protocol were also excluded.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Physical activity and constipation relationship | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Tantawy, PhD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Dr Dalia Kamel, Giza, Giza Governorate
  - Dr Sayed Tanatwy, Giza, Giza Governorate

IPD SHARING:
Plan to Share IPD: Yes
publication